CLINICAL TRIAL: NCT01517880
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Dose and Pharmacodynamic Efficacy of Sialic Acid-Extended Release (SA-ER) Tablets in Patients With GNE Myopathy or Hereditary Inclusion Body Myopathy
Brief Title: A Phase 2 Study to Evaluate the Dose and Pharmacodynamic Efficacy of Sialic Acid-Extended Release (SA-ER) Tablets in Patients With GNE Myopathy or Hereditary Inclusion Body Myopathy
Acronym: GNE Myopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UX001-CL201
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: GNE Myopathy; Hereditary Inclusion Body Myopathy
Keywords: Hereditary Inclusion Body Myopathy (HIBM); GNE myopathies; distal myopathy with rimmed vacuoles [DMRV]; Nonaka disease
MeSH Terms: conditions — Distal myopathy, Nonaka type

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 6,000 mg SA-ER (Experimental): Subjects will receive this dose for the duration of the study (total study duration of 48 weeks).
  Interventions: Drug: Sialic Acid Extended Release (SA-ER)
- Placebo (Placebo Comparator): Subjects will be randomized to the placebo arm for the first 24 weeks of the study. Then, subjects in this arm will be re-randomized into either the 3,000 mg per day or 6,000 mg per day arm for the remaining 24 weeks of the study (48 weeks total study duration).
  Interventions: Drug: Placebo
- 3,000 mg SA-ER (Experimental): Subjects will receive this dose for the duration of the study (total study duration of 48 weeks).
  Interventions: Drug: Sialic Acid Extended Release (SA-ER)

INTERVENTIONS:
Drug: Sialic Acid Extended Release (SA-ER) — SA-ER will be administered in doses of 3000mg per day or 6000mg per day
  Arms: 3,000 mg SA-ER; 6,000 mg SA-ER
Drug: Placebo — Subjects will be randomized to the placebo arm for the first 24 weeks of the study. Then, subjects in this arm will be re-randomized into either the 3,000 mg per day or 6,000 mg per day arm for the remaining 24 weeks of the study (total study duration 48 weeks).
  Arms: Placebo

SUMMARY:
GNE myopathy or hereditary inclusion body myopathy (HIBM) is a severe progressive metabolic myopathy caused by a defect in the biosynthetic pathway for sialic acid (SA).

DETAILED DESCRIPTION:
GNE myopathy or hereditary inclusion body myopathy (HIBM) is a severe progressive metabolic myopathy caused by a defect in the biosynthetic pathway for sialic acid (SA). Substrate replacement therapy is a potential therapeutic strategy based on the success of replacing missing SA and reducing muscle disease in a relevant mouse model of the human disease (Malicdan et al., 2009). Successful use of SA replacement therapy in humans is believed to depend upon providing steady long-term exposure to the compound in an extended release form (such as Sialic Acid-Extended Release [SA-ER]), given SA's short half-life. Following a Phase 1 study to establish the pharmacokinetics (PK) for SA-ER, Ultragenyx is conducting this study to assess the dose and potential pharmacodynamic effect of restoring sialylation of muscle by treatment with SA-ER at two dose levels as compared to placebo when administered over two 24 week periods of time. The study will also evaluate safety, as well as the effect of SA-ER on clinical measures of muscle strength, mobility, function and self-reported disability and quality of life. Effects on muscle volume/mass and function and on serum biomarkers will be evaluated as exploratory measures. These data should allow the selection of a dose and the appropriate design for a Phase 3 clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between 18 and 65 years of age, inclusive.
2. Must be willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
3. Must have a documented diagnosis of GNE myopathy, HIBM, distal myopathy with rimmed vacuoles (DMRV), or Nonaka disease due to previously demonstrated mutations in the gene encoding the GNE/MNK enzyme. Genotyping will not be conducted in this protocol.
4. Must be able to walk 20 meters independently (may use orthotics and assistive devices).
5. Must be able to provide reproducible force in bilateral elbow flexors and knee extensors during hand-held dynamometry testing (unilateral between test variability of < 15% for both muscle groups).
6. Must be willing and able to comply with all study procedures including fine needle muscle biopsies of the upper (e.g., triceps brachii or posterior deltoid) and lower (e.g., biceps femoris or vastus lateralis) extremities at Baseline and 24 and 48 weeks.
7. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
8. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause for at least two years, or have had tubal ligation at least one year prior to Screening, or who have had total hysterectomy.

Exclusion Criteria:

1. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.
2. Use of any investigational product or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
3. Ingestion of N-acetyl-D-mannosamine (ManNAc), SA, or related metabolites; intravenous immune globulin (IVIG); or anything that can be metabolized to produce SA in the body for the prior 60 days.
4. Has a condition of such severity and acuity, in the opinion of the investigator, that it warrants immediate surgical intervention or other treatment or may not allow safe participation in the study.
5. Has had any hypersensitivity to SA or its excipients that, in the judgment of the investigator, places the subject at increased risk for adverse effects.
6. Has a concurrent disease or condition that, in the view of the principal investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or would affect safety.
7. Has serum transaminase (i.e., alanine aminotransferase [ALT], aspartate aminotransferase [AST], or gamma-glutamyl transpeptidase [GGT]) levels greater than three times the upper limit of normal or serum creatinine of greater than 2.0 mg/dL.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of SA-ER treatment on muscle sialylation, strength, and function in patients with HIBM. | Baseline, Week 24, and Week 48
  To evaluate the effect of SA-ER treatment on improvement of biochemical measures of sialylation and pathology in muscle. On mobility, strength, and function using a series of quantitative and physical performance measures and quality of life using patient-reported outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Pestronk, MD, Principal Investigator — Washington University School of Medicine; Perry Shieh, MD, Principal Investigator — University of California, Los Angeles; Yoseph Caraco, MD, Principal Investigator — Hadassah University Hospital; Heather Lau, MD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (3):
  - UCLA Medical Center, Los Angeles, California
  - Washington University School of Medicine, St Louis, Missouri
  - New York University School of Medicine, New York, New York
- Hadassah University Hospital, Jerusalem, Israel